CLINICAL TRIAL: NCT05559996
Title: Assessment of the Efficacy of Multifractional Intercalated Hyaluronic Acid Injection for Genitourinary Syndrome of Menopause
Brief Title: Assessment of the Efficacy of Injectable Hyaluronic Acid for Genitourinary Syndrome of Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/900/88
Record Dates: First submitted 2022-09-22; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: vulvovaginal atrophy; hyaluronic acid; menopause; sexual dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyaluronic acid injection (Experimental): Hyaluronic acid injection
  Interventions: Device: Injectable form of multifractional intercalated cross-linked hyaluronic acid (Armonia®, Regenyal, Italy)

INTERVENTIONS:
Device: Injectable form of multifractional intercalated cross-linked hyaluronic acid (Armonia®, Regenyal, Italy) — 2 mL of Armonia was injected into the vaginal wall with a standardized injection technique called Cannulated Intravaginal Injection Technique®. In this technique, Armonia® was injected as drops at 40 different points on the entire vaginal wall using 8 different entry points

SUMMARY:
The vaginal wall consists of epithelium, lamina propria, muscularis and adventitia (1). The decrease in postmenopausal estrogen levels causes thinning of the vaginal wall thickness and the development of genitourinary menopause syndrome (GSM), which is characterized by vaginal dryness, burning, pruritus, urinary complaints and sexual discomfort (2).

In the treatment of GSM symptomatology, there are many different non-hormonal treatment options such as vaginal topical agents and energy-based devices, as well as estrogen-based hormonal therapies (3). The main problem with non-hormonal treatments is the short-term resolution of vaginal atrophy and the lack of long-term results, while contraindications such as breast cancer history and unwillingness of the women to use hormones are problematic for estrogen-based treatments.

Considering all these issues, there is a search for new therapeutic agents with long and high efficiency and safety profile in the treatment of GSM. Hyaluronic acid (HA) which is one of the main components of the extracellular matrix and has water-binding property that provides moisturizing and lubricating effect (4). Besides, it is also reported as the key to the process of tissue regeneration through inflammation, cellular migration and angiogenesis (5). For these reasons, it seems to be a promising treatment of GSM symptomatology.

HA has many routes of administration, such as vaginal gels, ovules, and suppositories, and studies have shown that locally applied HA preparations have a short-term therapeutic effect on GSM symptoms (6). However, there is no consensus regarding HA efficacy due to heterogeneity of studies. Since it is an endogenous molecule, it can be thought that it will be more effective if it is injected directly into the epithelium rather than locally applied.

The injectable form of multifractional intercalated cross-linked HA (MIC-HA) (Armonia®, Regenyal, Italy) is designed for the reinforcement of the extracellular matrix in the female genital area. We intend to investigate and objectively evaluate the efficacy of MIC-HA injection on GSM symptoms and sexual functions in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

Vaginal dryness Burning Itching Dyspareunia Genital discomfort

-

Exclusion Criteria:

Presence of pelvic organ prolapse Vaginal infections History of genital carcinoma Vulvovaginal dystrophic diseases Previous vaginal surgery Current use of vaginal moisturizer or lubricant, and use of estrogen History of allergies to hyaluronic acid, betadine or lidocaine

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
vaginal punch biopsy | One month
  4-6 millimeter depth vaginal punch biopsy was taken from the posterior wall of vagina, between 6 and 7 o'clock, 1 cm inside from the hymen by a true-cut punch biopsy device (Robbins® True-Cut Disposable Biopsy Punch 5mm, Robbins Instruments, 2003 Edwards St. Houston, TX 77007). Histologically, epithelial thickness, vascularity and dermal papilla prominence were evaluated. Periodic acid schiff (PAS) staining was used to evaluate glycogenization in epithelial cells, while Masson's trichrome histochemical staining was used to evaluate the distribution and density of collagen (neo-collagenization) in the lamina propria

SECONDARY OUTCOMES:
Turkish validated form of the Female Sexual Function Index | One month
  2 (minimum)-36 (maximum). Higher scores mean better outcome

OTHER OUTCOMES:
Visual Analog Scale | One month
  0 (minimum)-10 (maximum). Higher scores mean worse outcome
Vaginal health index score | One month
  5 (minimum)-25 (maximum). Higher scores mean better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University Faculty of Medicine, Istanbul, Turkey (Türkiye)